CLINICAL TRIAL: NCT01403454
Title: Web-based IHCA for Successful Home Dialysis
Brief Title: Web-based Interactive Health Communication Application (IHCA) for Successful Home Dialysis
Acronym: WISHED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Scott Brimble, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-3536; Grant (Other Grant/Funding Number: AHSC AFP Innovation Fund)
Record Dates: First submitted 2011-07-21; First posted 2011-07-27 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; web-based application; dialysis education
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- usual care (No Intervention)
- Health Communication Application (Active Comparator)
  Interventions: Behavioral: Interactive Health Communication Application

INTERVENTIONS:
Behavioral: Interactive Health Communication Application — web-based application
  Arms: Health Communication Application

SUMMARY:
This study involves Chronic Kidney Disease patients that must choose the type of dialysis therapy they ultimately wish to perform. These patients receive education regarding dialysis types from nurses and Nephrologists at a Kidney Function Program. The investigators have developed a web-based Interactive Health Communication Application that could provide more education and support to patients about their dialysis choices. The investigators will compare patients that will receive usual care dialysis education versus patients that will receive additional education through this web-based application. The investigators feel that this tool may increase the proportion of patients who start home dialysis, which offers advantages such as improvement in quality of life and deceased overall healthcare costs, over hospital hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in Kidney Function Program (KFP)
* previously received KFP-administered dialysis modality education
* personal access to a home computer (ie. either their own or a close friend/family member) with internet access
* most recent eGFR < or = 20mL/min/1.73m2

Exclusion Criteria:

* inability to provide informed consent
* inability to use a home computer or internet
* inability to understand English (written or spoke)
* severe visual or auditory impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients that start home-based dialysis. | 1 year
  Difference between groups in proportion of patients starting home-based dialysis.

SECONDARY OUTCOMES:
Number intended to start home-based dialysis | 1 year
  Difference between groups in proportion of patients intending to perform home-based dialysis
Increase in dialysis knowledge | 1 year
  Difference between groups in dialysis knowledge.
Increase in decision making and social support. | 1 year
  Difference between groups in decision conflict and sense of social support.
Mortality differences | 1 year
  Difference between groups in all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Scott K Brimble, MD, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Molnar AO, Harvey A, Walsh M, Jain AK, Bosch E, Brimble KS. The WISHED Randomized Controlled Trial: Impact of an Interactive Health Communication Application on Home Dialysis Use in People With Chronic Kidney Disease. Can J Kidney Health Dis. 2021 Jun 4;8:20543581211019631. doi: 10.1177/20543581211019631. eCollection 2021. PMID 34158965
- [Derived] Harvey A, Walsh M, Jain AK, Bosch E, Moreau C, Garland J, Brimble KS. The WISHED Trial: implementation of an interactive health communication application for patients with chronic kidney disease. Can J Kidney Health Dis. 2016 Jun 15;3:29. doi: 10.1186/s40697-016-0120-y. eCollection 2016. PMID 27307996